CLINICAL TRIAL: NCT00005608
Title: Orzel (UFT+Leucovorin) as First-Line Therapy for Metastatic Breast Cancer
Brief Title: Fluorouracil-Uracil and Leucovorin in Treating Women With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug was pulled from the market.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 99B3; NU-99B3; BMS-NU-99B3; NU-DRUG-BMS-ORZEL; NCI-G00-1741
Record Dates: First submitted 2000-05-02; First posted 2004-04-19 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Leucovorin; Tegafur

INTERVENTIONS:
Drug: leucovorin calcium
Drug: tegafur-uracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of fluorouracil-uracil and leucovorin in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate in women with metastatic breast cancer treated with fluorouracil-uracil and leucovorin calcium as first line therapy. II. Determine time to disease progression in this patient population treated with this regimen. III. Evaluate the toxicity profile of this regimen in these patients.

OUTLINE: Patients receive oral fluorouracil-uracil and oral leucovorin calcium twice daily for 28 days followed by 1 week of rest. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression. Patients with responding disease receive a minimum of 6 courses of treatment. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 22-33 patients will be accrued for this study within 13-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Metastatic breast cancer Bidimensionally measurable or evaluable disease No bone metastases as only site of measurable or evaluable disease that has been receiving bisphosphonate therapy for less than 2 months No known evidence of brain metastases, lymphangitis lung metastases, or carcinomatous meningitis Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: ECOG 0-1 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST or ALT no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Calcium no greater than 1.3 times ULN Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No history of other cancers except curatively treated carcinoma in situ of the cervix or nonmelanomatous skin cancer No active serious infection or other serious underlying medical condition that would preclude study therapy No dementia or significantly altered mental status that would preclude study consent No known hypersensitivity to fluorouracil-uracil or leucovorin calcium

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Concurrent colony stimulating factors (e.g., filgrastim (G-CSF), sargramostim (GM-CSF)) allowed only during time off treatment during each course Chemotherapy: No prior chemotherapy for metastatic disease At least 6 months since prior adjuvant chemotherapy and recovered Prior adjuvant fluorouracil allowed provided not infusional No prior fluorouracil-uracil with or without leucovorin calcium, capecitabine, S-1, or ethynyl uracil No other concurrent chemotherapy Endocrine therapy: Prior hormonal therapy for metastatic disease or in adjuvant setting allowed Recovered from toxicity No concurrent hormonal anticancer therapy Radiotherapy: Prior radiotherapy for metastatic disease or in adjuvant setting allowed At least 2 weeks since prior radiotherapy and recovered No prior radiotherapy to greater than 30% of bone marrow No concurrent radiotherapy except for palliation of painful bone metastases, pathologic fractures of known lytic disease, or brain lesions that develop Surgery: Not specified Other: No other concurrent investigational therapy No other concurrent anticancer drugs No concurrent halogenated antiviral agents (e.g., lodenosine, fialuridine, L-FMAU, emtricitabine, or sorivudine) No concurrent initiation of bisphosphonate therapy for development of new bone lesions or progression of existing bone lesions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States